CLINICAL TRIAL: NCT00636558
Title: A Phase I, Open-Label, Cohort Study of Multiple Doses of Cavatak™ (Coxsackie Virus A21) Given Intravenously to Stage IV Solid Tumour Cancer Patients Bearing ICAM-1 With or Without DAF Expressing Tumours (PSX-X04)
Brief Title: Coxsackie Virus A21 Administered Intravenously (IV) for Solid Tumour Cancers (PSX-X04)
Acronym: PSX-X04
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-004; PSX-X04 (Other: Viralytics Study ID)
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Melanoma; Breast Cancer; Prostate Cancer
Keywords: coxsackie virus; melanoma; breast cancer; prostate cancer
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Prostatic Neoplasms; Coxsackievirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CVA21 (Experimental): IV administration of CVA21 in a dose escalation manner
  Interventions: Drug: CVA21

INTERVENTIONS:
Drug: CVA21 — IV infusion, dose escalation of one or two infusions of escalating strength
  Other Names: CAVATAK

SUMMARY:
Coxsackie A21 (CVA21) virus is to be administered by IV infusion to patients with Stage 4 melanoma, prostate and breast cancer. This is a dose escalation, safety study.

DETAILED DESCRIPTION:
This is a phase I, multiple dose, dose escalation, open label, cohort study of three intravenous doses of Coxsackie virus A21 in patients with stage IV solid tumours. Prospective patients will attend the study centre for initial screening within 28 days prior to commencement of treatment. They will have the nature of the study and its procedures and risks fully explained. Patients must then sign an informed consent form giving permission for tumour testing before initial screening can be commenced.

Patients whose tumours test positive for ICAM-1 with or without DAF will attend the study centre for a further screening visit within 14 days prior to commencement of treatment. They will sign a full study informed consent form before any further screening procedures are carried out.

Patients who satisfy all inclusion and none of the exclusion criteria will commence the treatment stage, which consists of one or more doses of CVA21 administered by intravenous infusion as per the dosage escalation chart. The first 4 cohorts will be treated as in-patients. The follow up period will consist of 12 weeks, during which time patients will attend the trial centre for up to13 follow up visits to collect safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing and able to provide written informed consent to participate in the study.
2. Male or female aged 18 years or older.
3. Stage IV solid tumour disease with the primary tumour being any one of the following types - breast, prostate or melanoma.
4. ICAM-1 with or without DAF-expressing tumour. Patients without archival material for testing must agree to a new tumour biopsy.
5. Absence of circulating antibodies to CVA21 (titre < 1:16).
6. Patients must have failed or refused standard treatment(s).
7. Adequate haematological, hepatic and renal function, defined as:

   * ANC > 1.5 x 10^9/L, platelets > 100 x 10^9/L
   * Bilirubin < 20µmol/L, AST < 2.5 times the upper limit of normal
   * Calculated creatinine clearance > 30 mL/minute
8. Adequate immunologic function, defined as:

   * Serum IgG > 5g/L
   * T cell subsets within normal limits
9. Fertile males and females must agree to the use of an adequate form of contraception. Hormonal contraceptives should be supplemented with an additional barrier method. Negative pregnancy test is required in female patients of child-bearing potential.

Exclusion Criteria:

1. Presence or history of Central Nervous System (CNS) malignancy.
2. Patients must not have received chemotherapy within 4 weeks prior to date of consent.
3. Performance status > 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
4. Life expectancy < 6 months.
5. Pregnancy or breastfeeding.
6. Primary or secondary immunodeficiency, including immunosuppressive disease, and immunosuppressive doses of corticosteroids (e.g. prednisolone > 7.5mg per day) or other immunosuppressive medications including cyclosporine, azathioprine, interferons, within the past 4 weeks.
7. Positive serology for HIV, hepatitis B or hepatitis C.
8. Splenectomy.
9. Presence of uncontrolled infection.
10. Presence of unstable neurological disease.
11. Any uncontrolled medical condition that in the opinion of the Investigator is likely to place the patient at unacceptable risk during the study or reduce their ability to complete the study
12. Participation in another study requiring administration of an investigational drug or biological agent within the last 4 weeks
13. Known allergy to treatment medication or its excipients
14. Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2012-01-12 (Actual); Study Completion 2012-01-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to determine the safety and tolerability of CVA21 given by intravenous infusion in multiple escalating doses. | Days 1, 2, 5, 6, 7, 8, 12, 16, 20, 28, 42, 56, 84

SECONDARY OUTCOMES:
To obtain preliminary efficacy data, determine the time course of viraemia and its elimination post-administration of CVA21 | Days 1, 2, 5, 6, 7, 8, 12, 16, 20, 28, 42, 56, 84
To characterise the time course of the anti-CVA21 antibody response | Days 1, 2, 5, 6, 7, 8, 12, 16, 20, 28, 42, 56, 84

CONTACTS AND LOCATIONS:
Overall Officials: Boris Chern, MD, Principal Investigator — Redcliffe Hospital, Brisbane, Qld., Australia; Winston Liauw, MD, Principal Investigator — St George Hospital
Locations (2):
- Australia (2):
  - Cancer Care Centre, St George Hospital, Kogarah, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland